CLINICAL TRIAL: NCT02762214
Title: Role Of Uterine Manipulator in Hysterectomy for Early Stage Endometrial Cancer
Brief Title: Role of Uterine Manipulator in Hysterectomy - Ro.Man.HY
Acronym: RoManHy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RoManHy
Record Dates: First submitted 2016-04-16; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Endometrial Cancer
Keywords: Uterin manipulator; Endometrial Cancer; Laparoscopy; Robotic
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Uterine Manipulator (Active Comparator): 77 Patients affected by early stage endometrial cancer submitted to elective laparoscopic/robotic hysterectomy for endometrial cancer using uterine manipulator.
  Interventions: Device: Clermont-Ferrand Uterine Manipulator
- Without Uterine Manipulator (Experimental): 77 Patients affected by early stage endometrial cancer submitted to elective laparoscopic/robotic hysterectomy for endometrial cancer without support of uterine manipulator.
  Interventions: Other: No uterine Manipulator

INTERVENTIONS:
Device: Clermont-Ferrand Uterine Manipulator — Pelvic cytology is obtained before starting surgical procedures (washing number 1).
  After tubal coagulation, Clermont-Ferrand Uterine Manipulator is installed inside the uterus. At the end of the hysterectomy, after colporrhaphy, a second cytology is obtained (washing number 2)
  Arms: With Uterine Manipulator
Other: No uterine Manipulator — Pelvic cytology is obtained before starting surgical procedures (washing number 1). None uterine manipulator is used and the cervix is closed with a cross stitch.
  Tubal coagulation, At the end of the hysterectomy, after colporrhaphy, a second cytology is obtained (washing number 2)
  Arms: Without Uterine Manipulator

SUMMARY:
Prospective multicentric randomized trial to evaluate the role of uterine manipulator on laparoscopic/robotic total hysterectomy for the treatment of early stage G1 - G2 endometrial cancer (International Federation of Gynecology and Obstetrics - FIGO stages IA-IB).

DETAILED DESCRIPTION:
This multicentric prospective randomized Phase III trial is aimed to verify if the use of uterine manipulator for laparoscopic/robotic treatment of early stage endometrial cancer can influence the impact of peritoneal cytology and lymph vascular space invasion (LVSI) and the outcomes in terms of perioperative and oncological (disease free survival - DFS, overall survival - OS) outcomes.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Age > 18 < 80 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* No actual pregnancies
* Body Mass Index (BMI) ≤ 35

For diseases

* Early stage endometrial cancer (IA-IB)
* Endometrioid histotype (G1-G2)

Exclusion Criteria:

For patients

* Age > 18 < 80
* Actual pregnancies
* Previous gynecological cancer

For disease

* Type II endometrial cancer histotype
* Grade 3 endometrial cancer
* Advanced stage endometrial cancer (II - IV)
* Previous radiotherapy on the pelvic field
* Uterine size larger than conform 12 weeks gestation or 9 cm in horizontal
* Necessity of laparotomic procedures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Upstaging rate | 30 days
  Evaluation of Lymphovascular space invasion and pre- / post-Hysterectomy pelvic cytology in order to investigate if the use of uterine manipulator has a role in upstaging of early-stage endometrial cancer

SECONDARY OUTCOMES:
Complications | within 30 days from surgery
  To measure intra- and postoperative complication rate in order to investigate the specific role of uterine manipulator in complication occurred during hysterectomy or within 30 days after.
Blood Loss | Intraoperative
  To measure intraoperative estimated blood loss (EBL) in order to investigate the specific role of uterine manipulator in hemostatic control during Hysterectomy safety of laparoscopic hysterectomy
Impact of surgical procedure | Perioperative
  To measure the specific role of uterine manipulator in impact on surgery. More in dept operative time (OT), ileus, discharge time will be respectively measured in minutes, hours and days.
Role of uterine manipulator in Obesity | Intraoperative
  To determine the specific correlations between the use or not of uterine manipulator and Body Mass Index (BMI measured in kg/m2). To investigate if even this issue could influence the intraoperative safety
Impact on postoperative pain | Postoperative
  To investigate if the use or not of uterine manipulator could have a role in postoperative pain. Visual Analog Score (VAS) will be used to evaluate it.
Oncological Outcomes: Rate of local relapses | 1 years - 5 years
  To investigate if the use or not of uterine manipulator could determine an higher rate of local relapses

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Oncologic Gynecology, Fondazione Policlinico Gemelli, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided